CLINICAL TRIAL: NCT03976284
Title: Garden-fresh Produce and Exercise Reduce Colon Cancer Risk by Reducing Central Obesity and Increasing Stool Quality
Brief Title: Garden-fresh Produce and Exercise Reduce Colon Cancer Risk
Acronym: GFPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Charles Drew University of Medicine and Science (Other)
Responsible Party: Principal Investigator, William J. McCarthy, Ph.D., Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: U54CA14393009
Record Dates: First submitted 2019-06-01; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Garden-fresh Produce and Exercise (GFPE)
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will participate in 10 weekly health promotion sessions featuring cooking instruction, brief didactic nutrition instruction and 10-minute bouts of physical activity all taking place in the church kitchen/meeting room.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Garden-fresh produce and exercise (GFPE) (Experimental): Participants are encouraged to double their consumption of minimally processed fiber-rich plant foods, especially garden-fresh produce from the church community garden. Participants are also encouraged to limit pro-inflammatory foods rich in saturated fat, sodium and added sugar. Participants are also encouraged to engage in 150 minutes of moderate to vigorous physical activity per week, most likely in the form of brisk walking.
  Interventions: Behavioral: Garden-fresh produce and exercise

INTERVENTIONS:
Behavioral: Garden-fresh produce and exercise — The Garden-fresh produce and exercise (GFPE) health promotion intervention features 10 weekly sessions that take place after Sunday services in the Lincoln Memorial Church kitchen/meeting space. Each session includes a cooking demonstration focused on how to prepare and cook a meal composed of fiber-rich plant foods minimally processed. Each session also includes brief, didactic nutrition instruction and a 10-minute bout of physical activity.
  Other Names: GFPE

SUMMARY:
The investigators propose a church-based health promotion program designed to reduce colon cancer risk in a mostly African American community served by the Lincoln Memorial Church in South Los Angeles. The investigators propose involving 20 overweight/obese community members in a 10-session health promotion program featuring weekly cooking classes, didactic nutrition instruction and brief bouts of exercise. Behavioral aim is to increase participants' fiber intake from commonly consumed plant foods and reduce their intake of pro-inflammatory foods. They will be followed for 3 months from time of enrollment. Intervention is expected to increase participants' mean stool weight and improve their Bristol Stool Chart score. Intervention is expected to reduce waist circumference and systolic blood pressure of participants. These effects are expected to be accompanied by self-reports of increased fiber intake and reduced intake of saturated fat and refined sugar as well as evidence of increased physical activity.

DETAILED DESCRIPTION:
The investigators propose a church-based health promotion program designed to reduce colon cancer risk in a mostly African American community served by the Lincoln Memorial Church in South Los Angeles. The Los Angeles County of Public Health has divided the county into nine service planning areas (SPAs), of which South LA is one. Of all the SPAs, the South LA SPA has the highest prevalence of obesity and the lowest adherence to federal nutrition recommendations. With seed grant funds from a cooperative NIH grant shared by the Drew School of Medicine and University of California-Los Angeles (UCLA), the Lincoln Memorial Church of Los Angeles is sponsoring a behavioral intervention featuring 10 weekly sessions composed of cooking demonstrations, brief didactic nutrition education and 10-minute exercise bouts. All sessions will take place in the church kitchen and meeting room. Participants are expected to be 20 mostly African American, overweight/obese community members. The behavioral goal of the health promotion sessions is to encourage participants to eat more fiber-rich plant foods, minimally processed, to consume fewer pro-inflammatory foods including foods rich in saturated fat, sodium and refined sugar, and to engage in federally recommended amounts of physical activity. If research resources become available to enable blood chemistry results and/or fecal metagenomic results, the investigators would predict that 3 months after participant enrollment in the study, participants would experience a reduction in their high-sensitivity-C-reactive protein concentration and an increase in the relative abundance of obligate anaerobic bacteria relative to other bacteria in fecal samples. As seems likely, however, results will be limited to evaluating the weight and form of participant stool samples using the Bristol Stool Chart and evaluating participants' waist circumference and systolic blood pressure. The 3 month follow-up assessment is expected to show increased stool weight, improved Bristol Stool Chart score, decreased waist circumference, decreased systolic blood pressure, reduced intake of saturated fat and refined sugar, and increased weekly physical activity.

ELIGIBILITY:
Inclusion Criteria:

* body mass index > 25 > 40.
* must reside within 5 miles of the Lincoln Memorial Congregational Church
* must understand English

Exclusion Criteria:

* Crohns disease, ulcerative colitis or irritable bowel syndrome
* currently taking any prescription medication likely to cause weight gain or weight loss
* Currently taking medication for diabetes (e.g., metformin, insulin)
* Had a heart attack in the last 12 months
* Ever had bariatric surgery (weight loss surgery)
* Have been hospitalized for a mental health problem in the last 12 months
* Are currently pregnant or breastfeeding
* Currently use tobacco products such as cigarettes, electronic cigarettes
* Currently use marijuana products, including edibles

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-17 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Stool weight | At baseline and 3 months post-enrollment
  Mean stool weight of single bowel evacuation using precision digital scale

SECONDARY OUTCOMES:
Bristol Stool Chart score | At baseline and 3 months post-enrollment
  Bristol Stool Chart score ranges from 1 (hard lumps) to 7 (soft, diarrhea, liquid)
Waist circumference | At baseline and 3 months post-enrollment
  Waist circumference measured over light clothing using tensioner-equipped waist circumference measuring device
Systolic blood pressure | At baseline and 3 months post-enrollment
  Resting blood pressure assessed in participant seated quietly at a table with legs uncrossed
Ratio of fruit and vegetable fiber intake to total solid food intake | At baseline and 3 months post-enrollment
  The ratio of fruit and vegetable fiber intake relative to total gram weight of foods consumed per day based on data from Block Food Frequency questionnaire.
Saturated fat intake | At baseline and 3 months post-enrollment
  Mean grams (g) of saturated fat intake consumed daily based on retrospective food consumption data obtained from administration of the Block Food Frequency questionnaire. The Daily Value for saturated fat is less than 20 g per day, based on a 2,000 calorie diet. Meat-eating Americans generally consume more than 20 g per day but usually don't exceed 80 g per day. Humans make all the saturated fat that they need, so consuming zero g of saturated fat per day is consistent with good health.
Sugary beverage intake | At baseline and 3 months post-enrollment
  Percent of daily calorie intake attributable to sugary beverage intake

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Center for Cancer Prevention & Control Research, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Because the pilot study sample is small (N=20), the likelihood of deductive disclosure of identity is high even if the shared data were de-identified. Hence, there will be no sharing of individual level data with other researchers not originally comprising the investigative team.